CLINICAL TRIAL: NCT07144241
Title: Mesenchymal Stromal/Stem Cells-Derived Exosomes (MSC-Exos) Therapy for Type 2 Diabetes Mellitus Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Yanuar Ardani, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YArdani MSC-Exos T2DM
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: DMT2; Mesenchymal Stromal/Stem Cells-Derived Exosomes; Glycemic Profile; Quality of Life; Inflammatory Biomarkers
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: open-label randomized controlled trial with a pre-and-post-test control group design. The study aims to compare the effectiveness of Mesenchymal Stromal/Stem Cells-Derived Exosomes (MSC-Exos) as an additional therapy for patients with Type 2 Diabetes Mellitus (T2DM).
  The study will recruit 50 subjects who meet the inclusion and exclusion criteria. These subjects will be randomly assigned to one of two groups Intervention Group: This group will receive standard T2DM therapy along with a combination of exosomes, specifically 1 vial of Exo-HWS and 1 vial of Exo-HUVEC. The exosome therapy will be administered as an intravenous bolus injection monthly, for three months.
  Control Group: This group will receive standard T2DM therapy plus 1 vial of Exo-HWS. This therapy will also be administered monthly, for three months, via intravenous bolus injection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Intervention Group (Active Comparator): Receives standard therapy for Diabetes Mellitus (DM) plus a combination of exosomes (1 vial Exo-HWS + 1 vial Exo-HUVEC).
  Administered as a monthly intravenous bolus injection for three months
  Interventions: Biological: Mesenchymal Stromal/Stem Cells-Derived Exosomes (Exo-HWS + 1 vial Exo-HUVEC) Therapy
- Group 2: Control Group (Placebo Comparator): Receives standard therapy for DM plus 1 vial of Exo-HWS.
  Administered as a monthly intravenous bolus injection for three months.
  Interventions: Biological: Mesenchymal Stromal/Stem Cells-Derived Exosomes (Exo-HWS ) Therapy

INTERVENTIONS:
Biological: Mesenchymal Stromal/Stem Cells-Derived Exosomes (Exo-HWS + 1 vial Exo-HUVEC) Therapy — The intervention group will receive standard DM therapy plus an exosome combination of 1 vial Exo-HWS + 1 vial Exo-HUVEC, administered monthly for three months via intravenous bolus injection.
  Arms: Group 1: Intervention Group
Biological: Mesenchymal Stromal/Stem Cells-Derived Exosomes (Exo-HWS ) Therapy — The control group will receive standard DM therapy plus 1 vial Exo-HWS, administered monthly for three months via intravenous bolus injection.
  Arms: Group 2: Control Group

SUMMARY:
This is an open-label randomized controlled trial with a pre-and-post-test control group design to evaluate the effect of Mesenchymal Stromal/Stem Cells-Derived Exosomes (MSC-Exos) as an adjunctive therapy on glycemic control and clinical outcomes in patients with Type 2 Diabetes Mellitus (T2DM). The study aims to determine if the addition of exosome therapy to standard care can improve glycemic parameters (fasting blood glucose, 2-hour postprandial glucose, HbA1c, and C-peptide), quality of life, and inflammatory biomarkers (IL-6, IL-10, D-dimer, and CRP). The study will involve 50 subjects, randomly allocated into two groups: an intervention group and a control group. The intervention group will receive standard T2DM therapy plus a combination of exosomes (1 vial Exo-HWS + 1 vial Exo-HUVEC). The control group will receive standard T2DM therapy plus 1 vial Exo-HWS. The study duration is from June to December 2025.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Type 2 Diabetes Mellitus.
* Patients aged 40 to 65 years.
* Patients who are willing to participate in the study and sign the informed consent form after receiving a detailed explanation of the research procedure.

Exclusion Criteria:

* Patients with severe comorbidities that could affect the immune response, such as autoimmune diseases, malignancies, and severe infections.
* Patients currently undergoing anticoagulant therapy.
* Patients currently undergoing immunosuppressive therapy.
* Pregnant women, as the effects of exosome therapy on them have not been sufficiently studied.
* Patients with a history of severe allergies to components of the exosome therapy.
* Patients with CKD (Chronic Kidney Disease) on HD (Hemodialysis).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Fasting Blood Glucose (FBG) | Baseline (Day 0) and End of the 3rd Month
  Change in FBG levels from baseline to the end of the third month. Unit of Measurement: mg/dL
2-Hour Postprandial Glucose | Baseline (Day 0) and End of the 3rd Month
  Change in 2-hour postprandial glucose levels from baseline to the end of the third month.
  Unit of Measurement: mg/dL
HbA1c | Baseline (Day 0) and End of the 3rd Month
  Change in HbA1c levels from baseline to the end of the third month. Unit of Measurement: %
C-peptide | Baseline (Day 0) and End of the 3rd Month
  Change in C-peptide levels from baseline to the end of the third month. Unit of Measurement: ng/m

SECONDARY OUTCOMES:
Quality of Life using DQoL | Baseline (Day 0) and End of the 3rd Month
  Change in quality of life scores as measured by the Diabetes Quality of Life (DQoL) questionnaire from baseline to the end of the third month.
  Unit of Measurement: Score
IL-6 | Baseline (Day 0) and End of the 3rd Month
  Change in Interleukin-6 (IL-6) levels from baseline to the end of the third month.
  Unit of Measurement: mg/L
IL-10 | Baseline (Day 0) and End of the 3rd Month
  Change in Interleukin-10 (IL-10) levels from baseline to the end of the third month.
  Unit of Measurement: mg/L
D-dimer | Baseline (Day 0) and End of the 3rd Month
  Change in D-dimer levels from baseline to the end of the third month. Unit of Measurement: ng/mL
CRP | Baseline (Day 0) and End of the 3rd Month
  Change in C-Reactive Protein (CRP) levels from baseline to the end of the third month.
  Unit of Measurement: mg/L

CONTACTS AND LOCATIONS:
Locations (1):
- UNIMUS Hospital, Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
There is no explicit plan to share Individual Participant Data (IPD) from this study. The research team's commitment to participant confidentiality is paramount. The informed consent form assures participants that their data and information will be kept confidential and will be used solely for the purpose of the research, education, and scientific development, without disclosing their identity. This approach aligns with the ethical clearance obtained for the study, which emphasizes protecting participant identity.

REFERENCES:
- [Background] Li CJ, Xiao Y, Sun YC, He WZ, Liu L, Huang M, He C, Huang M, Chen KX, Hou J, Feng X, Su T, Guo Q, Huang Y, Peng H, Yang M, Liu GH, Luo XH. Senescent immune cells release grancalcin to promote skeletal aging. Cell Metab. 2021 Oct 5;33(10):1957-1973.e6. doi: 10.1016/j.cmet.2021.08.009. Epub 2021 Sep 9. PMID 34614408
- [Background] Kalluri R, LeBleu VS. The biology, function, and biomedical applications of exosomes. Science. 2020 Feb 7;367(6478):eaau6977. doi: 10.1126/science.aau6977. PMID 32029601
- [Background] Lai RC, Yeo RW, Lim SK. Mesenchymal stem cell exosomes. Semin Cell Dev Biol. 2015 Apr;40:82-8. doi: 10.1016/j.semcdb.2015.03.001. Epub 2015 Mar 9. PMID 25765629
- [Background] Raposo G, Stoorvogel W. Extracellular vesicles: exosomes, microvesicles, and friends. J Cell Biol. 2013 Feb 18;200(4):373-83. doi: 10.1083/jcb.201211138. PMID 23420871
- [Background] American Diabetes Association. Standards of Medical Care in Diabetes-2021 Abridged for Primary Care Providers. Clin Diabetes. 2021 Jan;39(1):14-43. doi: 10.2337/cd21-as01. No abstract available. PMID 33551551
- [Background] Williams R, Karuranga S, Malanda B, Saeedi P, Basit A, Besancon S, Bommer C, Esteghamati A, Ogurtsova K, Zhang P, Colagiuri S. Global and regional estimates and projections of diabetes-related health expenditure: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2020 Apr;162:108072. doi: 10.1016/j.diabres.2020.108072. Epub 2020 Feb 13. PMID 32061820